CLINICAL TRIAL: NCT02765386
Title: Optimisation of Hybrid Fittings for Newly Implanted Cochlear Implant Recipients
Brief Title: Optimisation of Hybrid Fittings for Cochlear Implant Recipients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After several years of trying to recruit participants, it was decided to stop the study after recruiting only 12 participants.
Sponsor: The Hearing Cooperative Research Centre (Other)
Collaborators: Royal Victoria Eye and Ear Hospital (Other Government); Cochlear (Industry); University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC5610
Record Dates: First submitted 2016-04-14; First posted 2016-05-06 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Hearing Loss
Keywords: Cochlear implants; Hybrid fittings; Cross-over frequency
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cochlear Implant Recipients (Experimental): Newly implanted cochlear implant recipients with post-implantation acoustic hearing.
  Interventions: Device: Hybrid fittings for cochlear implant recipients

INTERVENTIONS:
Device: Hybrid fittings for cochlear implant recipients

SUMMARY:
When providing amplification post-implantation to residual acoustic hearing in the implanted ear, the lower frequency boundary can be modified to minimize or avoid overlap between the frequencies coded through acoustic hearing and those presented through electrical stimulation. This boundary is termed the cross-over frequency (Fc) and the effect of modifying this parameter will be investigated in this study. To avoid the research being confounded by prior bias for a particular frequency allocation, the study will be conducted with newly implanted recipients.

This study will also investigate whether tests which measure the ability to use low frequency hearing and objective measures can predict the preferred Fc and speech performance benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years of age)
2. Post-operative residual hearing in the implanted ear (defined as having an unaided threshold better than or equal to 80 dB HL at the 500 Hz frequency).
3. Implanted with the CI500 or CI24RE-series cochlear implants
4. User of the commercially available Nucleus 6 sound processor
5. User of the ACE strategy
6. Native speaker in the language used to assess speech perception performance
7. Willingness to participate in and to comply with all requirements of the protocol

Exclusion Criteria:

1. Additional handicaps that would prevent participation in evaluations
2. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the procedure and investigational device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Speech, Spatial and Qualities of Hearing (SSQ) scale | Testing at 18, 19, 22 and 25 weeks post-activation of cochlear implant
  Preference rating assessed using SSQ scale
Word recognition scores in quiet | Testing at 12, 15, 18, 19, 22 and 25 weeks post-activation of cochlear implant
  Open-set monosyllabic word scores in quiet
Speech recognition in noise | Testing at 12, 15, 18, 19, 22 and 25 weeks post-activation of cochlear implant
  Open-set speech recognition in noise

CONTACTS AND LOCATIONS:
Locations (1):
- The HEARing CRC, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No